CLINICAL TRIAL: NCT06125301
Title: The Multiple Sclerosis Self Monitoring Study: An Intervention Study on the Effect of Digital Self-monitoring-based Management of Relapsing and Remitting Multiple Sclerosis on Self-efficacy, Clinical Outcomes and Cost-effectiveness
Brief Title: Multiple Sclerosis Self Monitoring Study
Acronym: MSSM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Joep Killestein, Prof., Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NL75687.029.20
Record Dates: First submitted 2022-11-28; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Care as usual + weekly self-monitoring during one year follow-up and discussing app results with caregivers.
  Interventions: Device: MS Sherpa
- Control group (No Intervention): Care as usual.

INTERVENTIONS:
Device: MS Sherpa — MS sherpa® is a medical device, intended to support monitoring of persons with MS in order to give patients and their professional healthcare team(s) insight into the presence and progress of symptoms related to MS. MS sherpa® is a system consisting of a smartphone app for data collection and data presentation, a cloud service for data storage, analysis algorithms, and a clinician or research dashboard for user management and data visualization. The device measures the course of symptoms related to MS with respect to walking speed (average walking speed derived from the distance walked during a 2-minute walk), cognitive processing speed, number of correct answers on a smartphone variant of the symbol digit modalities test (SDMT) and patient reported outcomes, through predefined questionnaires regarding fatigue, amongst others. MS sherpa® measures changes in these parameters over time and shows these on an insights screen in the app and on the clinician dashboard.
  Arms: Intervention group

SUMMARY:
This study is a multicenter, prospective, randomized controlled trial (RCT) to compare the effectiveness of a smartphone-based self-monitoring and self-management tool on control self-efficacy with respect to standard clinical practice for patients with relapsing-remitting multiple sclerosis (RRMS). RRMS patients will be recruited and screened for study eligibility at four Dutch MS centers. Following inclusion, participants will be randomly allocated to the intervention group (use of MS sherpa® in addition to standard care) or control group (standard care only). The duration of follow-up is 12 months with study visits at baseline and 12 months, and additional study assessments coupled with every clinical visit as part of standard care during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form.
2. Able to comply with the study protocol, as judged by the investigator.
3. A minimum age of 18 years.
4. Have a definite diagnosis of RRMS according to the revised McDonald 2017 criteria.
5. Have a length of disease duration of ≥12 months, from date of MS diagnosis.
6. Have clinical disease activity (one or more reported relapses) and/or radiological disease activity (new/enlarged T2 lesions or T1 contrast-enhancing lesions) within the past 12 months.
7. Willing and able to install and use MS sherpa® on own smartphone with Android (version 4.4 or higher) or iOS (version 9 or higher) operating system.
8. Willing to stay for treatment with the same hospital during the year of study.
9. Willing to follow the rules of conduct as described in Appendix A during the year of study.

Exclusion Criteria:

1. EDSS of > 6.5 at baseline screening.
2. Presence of a cognitive, visual or upper extremity deficit that disables the use or measurements of MS sherpa® on the smartphone, as judged by the investigator.
3. Concomitant use of health monitoring apps or devices for MS during the study.
4. Concomitant participation in another intervention trial in MS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2024-08-15 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
the Multiple Sclerosis Self-Efficacy Control scale (MSSE-C) | One year
  the MS Self-Efficacy scale is an 18-item scale assessing self-rated certainty regarding specific behaviours related to functional independence and psychological management of MS. Items are rated on a scale from 10 (very uncertain) to 100 (very certain). The MSSE consist of two subscales by summing the respective items: SE Function, and SE Control.

SECONDARY OUTCOMES:
Decision making process - caregiver | One year
  Provider Decision Process Assessment Instrument (PDPAI) for neurologists, adapted with an additional five questions about the use of MS sherpa® in the decision-making process.
Decision making process - patient | One year
  Decisional Conflict Scale (DCS) for persons with MS, adapted with an additional five questions about the use of MS sherpa® in the decision-making process.

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, locatie VUmc, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No